CLINICAL TRIAL: NCT02342184
Title: Efficacy and Safety Study of GB-0998 for Guillain-Barré Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Blood Products Organization (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B211-13
Record Dates: First submitted 2014-12-25; First posted 2015-01-19 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-12

CONDITIONS: Guillain-Barré Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GB-0998 (Experimental)
  Interventions: Drug: GB-0998

INTERVENTIONS:
Drug: GB-0998
  Other Names: Venoglobulin-IH

SUMMARY:
This study will carry out to assess the efficacy of GB-0998 (intravenous immunoglobulin;400mg/kg/day for five days) in the treatment of the Guillain-Barré Syndrome based on the changes in Hughes Functional Grade (FG) as primary endpoint, and in addition, to assess the safety of GB-0998.

ELIGIBILITY:
Inclusion Criteria:

1. In principle, patients are able to receive the treatment within 2 weeks (with limits of 4 weeks) from the start of symptoms.
2. Patients with predominant motor neuropathy and FG is grade 4 or grade 5 (if symptoms is progressive, patients with FG is grade 3 involve in this study).
3. Patients with plasmapheresis, steroids and immune globulin therapy is no operation for this onset.

Exclusion Criteria:

1. Patients who have the anamnesis of shock or hypersensitivity to GB-0998.
2. Patients who have been diagnosed as hereditary fructose intolerance.
3. Patients who have impaired peripheral neuropathy except Guillain-Barré syndrome.
4. Patients with history of volatile organic solvent abuse, abnormal porphyrin metabolism, history of pharynx or cutaneous diphtheria, plumbism, poliomyelitis, botulism, hysterical paralysis, toxic neuropathy.
5. Patients who have received treatment of malignant tumors.
6. Patients who were administered immunoglobulin within 8 weeks before informed consent.
7. Patients who have been diagnosed IgA deficiency in their past history.
8. Patients with severe renal disorder or decreased cardiac function.
9. Patients who have the anamnesis of cerebro- or cardiovascular disorders, or symptom of these diseases.
10. Patients with high risk of thromboembolism.
11. Pregnant, lactating, and probably pregnant patients.
12. Patients who were administered other investigational drug within 12 weeks before consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with more than 1 grade improvement in Hughes Functional Grade (FG) | 4 weeks

SECONDARY OUTCOMES:
days required for 1 grade improvement of FG | 1,2,3,4,6,8,12 weeks
days required for 2 grade improvement of FG | 1,2,3,4,6,8,12 weeks
changes in FG | 1,2,3,4,6,8,12 weeks
proportion of patients with more than 1 grade improvement in the Arm Grade (AG) relative to baseline | 4weeks
days required for 1 grade improvement of the AG | 1,2,3,4,6,8,12 weeks
days required for 2 grade improvement of the AG | 1,2,3,4,6,8,12 weeks
changes in AG | 1,2,3,4,6,8,12 weeks
changes in grip strength | 1,2,4,8,12 weeks
changes in manual muscle testing (MMT) | 1,2,4,8,12 weeks
changes in activity of daily living (ADL) | 1,2,4,8,12 weeks
changes in motor nerve conduction velocity | 4,12 weeks
changes in FG on rescue treatment | 1,2,3,4,6,8,12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyoichi Nomura, Study Chair — Department of Neurology, Saitama Medical Center, Saitama Medical University, Saitama, Japan
Locations (1):
- Department of Neurology, Saitama Medical Center, Saitama Medical University, Kawagoe, Saitama, Japan